CLINICAL TRIAL: NCT03044093
Title: Mifepristone and Misoprostol Compared With Misoprostol Alone for Second Trimester Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0299-16-RMB
Record Dates: First submitted 2017-01-18; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Second Trimester Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MISOPROSTOL alone (Active Comparator): the common practice currently in our medical center for second trimester medical abortion/ Placebo
  Interventions: Drug: Placebo; Drug: Misoprostol
- Mifepristone and Misoprostol (Experimental): in addition to the common practice currently in our medical center for second trimester medical abortion we will add Mifepristone before administering Misoprostol.
  Mifepristone
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — The group that will get in addition to Misoprostol also Mifepristone
  Arms: Mifepristone and Misoprostol
Drug: Placebo — The group that will only get Misoprostol
  Arms: MISOPROSTOL alone
Drug: Misoprostol — Both groups will get think drug

SUMMARY:
Mifepristone and Misoprostol Compared With Misoprostol Alone for Second Trimester Abortion - a Double Blinded Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* healthy
* no allergy known to these drugs
* second trimester abortion

Exclusion Criteria:

* hematology diseases
* clotting factor deficiency

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hospital Stay Duration | Up to 24 months
  number of days of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No